CLINICAL TRIAL: NCT05448027
Title: Comparison Between the Low and High Intensity Laser Therapy in Young Females With Primary Dysmenorrhea
Brief Title: Low Versus High Intensity Laser Therapy on Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermine Ahmed Mohamed Ahmed El Labbad, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003428
Record Dates: First submitted 2022-02-06; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low intensity laser therapy group (Experimental): • Group (A): lt will include 26 participants suffering from primary dysmenorrhea who will receive low intensity laser therapy 3 sessions per cycle for 3 consecutive cycles (one session will be applied the day before menstruation and the other two sessions on the 1st and 2nd days of menstruation
  Interventions: Device: Low intensity laser therapy
- High intensity laser therapy group (Experimental): Group (B): It will include 26 participants suffering from primary dysmenorrhea who will receive high intensity laser therapy 3 sessions per cycle for 3 consecutive cycles (one session will be applied the day before menstruation and the other two sessions on the 1st and 2nd days of menstruation
  Interventions: Device: High intensity laser therapy

INTERVENTIONS:
Device: Low intensity laser therapy — It will be applied for Group (A), by a pulsed diode low intensity laser device (Endolaser 422 Cp 400, Enraf - nonius apparatus) (Enraf, Rootterdam, Netherlands). with a wave length of 905 nm, mean power output of 400 mWatt, frequency of 10000 Hz and dose of 300 J/cm² . Laser probe will be applied perpendicularly and directly with an irradiation time of 30 sec for each point
  Arms: Low intensity laser therapy group
Device: High intensity laser therapy — It will be applied for Group (B), by pulsed high intensity laser therapy with pulsed Nd:YAG laser produced by HIRO 3.0 devices (ASA, Arcugnano, Vicenza , Italy). The high intensity laser therapy apparatus used postulates (Nd:YAG), with pulsed emission of wave length ( 1064nm ), very high power peaks (3kW), high intensity obtained (up to 15,000 W/cm2), high level of fluency/energy density (510-1,780 mJ/cm), very short pulse duration (120-150 μs), low frequency (10-40 Hz), duty cycle of about 0.1 % and total energy of 880 J
  Arms: High intensity laser therapy group

SUMMARY:
Primary dysmenorrhea constitutes a significant health, social and economic problems. It involves a broad spectrum of both physical and emotional manifestations with a prevalence that can reach 50 up to 91 % in young women . Furthermore, it compromises the most common gynaecological alternations and the major cause of women academic and work absenteeism which obviously reduces quality of life, daily activities and economic situation due to decreased working hours.

NSAIDs are the first therapeutic line for primary dysmenorrhea; however, they might be accompanied by some undesirable side effects, such as dyspepsia, headache and drowsiness .

Laser treatment is non-invasive, painless, and can be easily administered in primary care settings for a wide range of conditions. Laser treatment significantly reduces pain level in both acute and chronic painful conditions by increasing the production of endorphins.

Low intensity laser therapy (LTTT) as a physical therapy modality with variety of therapeutic effects. There are various researches concluded that it is a safe therapeutic modality for the treatment of dysmenorrhea .

More recently, the pulsed neodymium-doped yttrium aluminum garnet (Nd:YAG) , a form of high-intensity laser therapy (HILT), was introduced to the field of physical therapy. The use of pulsed Nd:YAG lasers with high peak powers (3kW) and wave length of 1064 nm has been increasing and is considered as a non painful and non invasive modality that can stimulate areas that can't be reached with the low power lasers with patients reporting more significant pain reduction . Studies have documented the anti-inflammatory, anti-edematous, and analgesic effects of Nd:YAG lasers, justifying their use in patients with pain issues .

In fact, the HILT program is effective and has a more prolonged effect in pain reduction, and improving QOL with effects lasting up to 12 weeks post-treatment .

There is limited literature regarding the clinical results of high intensity laser treatment for primary dysmenorrhea , this may be contributed to its high cost. So, this research is an attempt to add to the clinical knowledge in this field as it will investigate the difference between the effect of low and high intensity laser therapy on primary dysmenorrhea with the quality of life improvement being the main point of concern .

DETAILED DESCRIPTION:
This study will be conducted on fifty two participants suffering from primary dysmenorrhea selected from Cairo Specialised Hospital( Department of Obestetrics and Gynaecology).

All females will be randomly divided into two equal groups:

* Group (A): lt will include 26 participants suffering from primary dysmenorrhea who will receive low intensity laser therapy 3 sessions per cycle for 3 consecutive cycles (one session will be applied the day before menstruation and the other two sessions on the 1st and 2nd days of menstruation).
* Group (B): It will include 26 participants suffering from primary dysmenorrhea who will receive high intensity laser therapy 3 sessions per cycle for 3 consecutive cycles (one session will be applied the day before menstruation and the other two sessions on the 1st and 2nd days of menstruation ).

All females will be given a full explanation of the study protocol and a consent form will be signed by each female before entry in this study

ELIGIBILITY:
Inclusion Criteria:

- A)

* All females will be clinically diagnosed by gynaecologist with primary dysmenorrhea .
* Score ≥ 50 or moderate on Menstrual Distress questionnaire (MDQ)
* Their ages will range from 18-25 years old.
* Their BMI will be less than 30 kg/m² (El-Kosery et al., 2020).
* Being virgin.
* Having regular menstruation for the last 6 months (every 28-30 days with no intermittent bleeding).

Voluntary acceptance to participate in the study

Exclusion Criteria:

* Participants will be excluded if they have :

  * Systematic chronic diseases , adenomyosis, pelvic inflammatory disease.. etc
  * Mental disability .
  * Professional athletes (Jill et al., 2012).
  * Secondary dysmenorrhea pathology.
  * Menstrual irregularity.
  * Using hormonal contraception (such as contraceptives and injections) .
  * Epileptic fits .
  * Cardiac pacemakers.
  * Lumbar disc lesions .

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 3 months
  It will be measured using visual analogue scale (VAS): It will be used to measure pain intensity for each female in both groups (A&B) . The VAS is usually presented as a 10 cm horizontal line on which the participants' pain intensity is represented by a point between the extremes of " no pain at all " and " worst pain imaginable ". It's simplicity , reliability and validity as well as its ratio scale properties make the VAS the optional tool for describing pain intensity
Menstrual symptoms | 3 months
  It will be assessed by Menstrual Distress questionnaire (MDQ): It consists of symptoms or feelings associated with menstruation. The total number of items is 47 . It is a 5 point rating scale from 0-4 . For each items , there is 5 options i.e. No, mild , moderate, severe and very severe . An option of (very severe) has a score of 4, (severe) has a score of 3, (moderate) has a score of 2, (mild) has a score of 1, (No) has a score of 0 . It includes seven subscales as (pain, water retention, autonomic reactions, negative affect, impaired concentration, mood and behavioral changes, arousal control). Overall Score was interpreted as follows:
  <50 - mild , 50 to 70 - moderate and >70 severe
Quality of life improvement | 3 months treatment and 3 months follow up
  It will be assessed by Quality of life enjoyment and satisfaction questionnaire Q-LES-QSF: It consists of items that evaluate overall enjoyment and satisfaction regarding ; Physical Health, mood, work, household and leisure activities, family and social relationships, ability to function in daily life , economic status , living or housing situation , ability to get around physically, ability to do work or hobbies, and overall sense of being. The Q-LES-Q-SF is a validated, self-reported evaluation of the degree to which enjoyment and satisfaction are derived from various areas of life
Pressure pain threshold | Pre and post treatment program I.e up to 3 months
  Pressure algometer: It is a device used to identify the pressure and / or force eliciting a pressure-pain threshold (PPT) . PPT occurs at the minimum transition point when applied pressure ( i.e. force) is sensed as pain . It is non- invasive, efficient and reliable tool in the exploration of physio-pathological mechanisms involved in muscle pain syndromesq